CLINICAL TRIAL: NCT06639204
Title: Evaluation of the Skeletal, Dental and Soft-tissue Changes After En-masse Retraction of the Upper Anterior Teeth Stimulated by Low-intensity Electrical Current: A Single-centered, Randomized Controlled Clinical Trial
Brief Title: Cephalometric Changes Following Retraction of the Upper Anterior Teeth Stimulated by Low-intensity Electrical Current
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-5-2024
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Class II Division 1 Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — Electric Stimulation; Orthodontics; Acceleration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrical Stimulation (Experimental): Electric current will be applied in this group of patients using a removable device.
  Interventions: Device: Electrical stimulation
- Conventional treatment with no stimulation (Active Comparator): No acceleration method will be performed in this group
  Interventions: Procedure: Orthodontic treatment without acceleration

INTERVENTIONS:
Device: Electrical stimulation — A removable appliance will be used to accelerate orthodontic tooth movement by emitting electrical stimulation.
  Arms: Electrical Stimulation
Procedure: Orthodontic treatment without acceleration — No additional appliances will be used. Only the traditional fixed appliances (braces).
  Arms: Conventional treatment with no stimulation

SUMMARY:
Thirty-six patients requiring extraction of maxillary first premolars and en-masse retraction of upper anterior teeth will participate in the study. They will be randomly assigned into two groups: low-intensity electrical stimulation group (LIES) and traditional retraction group (TRAD) after the leveling and alignment phase is completed. En-masse retraction will be initiated in both groups via closed nickel-titanium coil springs that applying 250 g of force on each side, Mini-implants will be inserted to provide the highest level of anchorage. The skeletal, dental, and soft tissue changes will be detected using lateral cephalometric radiographs, which will be obtained pretreatment, pre-, and post-en-masse retraction of the anterior teeth.

DETAILED DESCRIPTION:
All candidate patients will be examined to determine the orthodontic treatment plan. Written informed consent will be obtained from all patients who accept to participate in the trial. Self-drilling mini-screws (1.6mm diameter and 8mm length) will be used to provide anchorage. They will be inserted bilaterally 8-10 mm above the level of the interdental papilla, between the second premolars and the first molar. Then, the maxillary first premolar will be extracted. Leveling and alignment of the upper dental arch will be done using a pre-adjusted orthodontic appliance: MBT™, 0.022 × 0.028-inch slots-size brackets. The removable electrical stimulation device utilized in the Shaadouh et al. study to provide the electrical stimulation will be used in this trial for the same purpose. Each patient in the low-intensity electrical stimulation group will be asked to wear a removable device for five hours daily until the completion of the retraction of the upper anterior teeth.

The en-masse retraction will be done by applying 250 g force on each side using two NiTi springs attached between the mini-implants and the crimpable hooks in a direction approximately parallel to the occlusal plane. The force will be calibrated every two weeks. The en-masse retraction will continue until a class I canine relationship and a correct incisor relationship, which will consider the endpoint of this phase.

Lateral cephalometric radiographs will be obtained pretreatment, pre-, and post-en-masse retraction of the anterior teeth to assess the skeletal, dental, and soft tissue changes. The duration of retraction will be calculated by calculating the time required to achieve complete retraction of the upper anterior teeth through clinical examination.

ELIGIBILITY:
Inclusion Criteria:

1. Adult healthy patients, Male and female, Aged 18-25 years.
2. Class II Division 1 malocclusion :

   * Mild/moderate skeletal Class II (ANB= 5-7 degrees)
   * Overjet ≤10
   * Normal or excessive facial height (Clinically and then cephalometrically assessed using these three angles: mandibular/cranial base angle, maxillary/mandibular plane angle, and facial axis angle)
   * Mild to moderate crowding ≤ 4
3. Permanent occlusion.
4. Existence of all the upper teeth (except third molars).
5. Good oral and periodontal health:

   * Probing depth < 4 mm
   * No radiographic evidence of bone loss.
   * Gingival index ≤ 1
   * Plaque index ≤ 1

Exclusion Criteria:

1. Medical problems that affect tooth movement (corticosteroids, nonsteroidal anti-inflammatory drugs (NSAIDs), …)
2. Presence of primary teeth in the maxillary arch
3. Missing permanent maxillary teeth (except third molars).
4. Poor oral hygiene or Current periodontal disease:

   Probing depth ≥ 4 mm Radiographic evidence of bone loss Gingival index > 1 Plaque index > 1
5. Patient had previous orthodontic treatment

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Duration of the en-masse retraction of anterior teeth | At the end of en-masse retraction which is expected to occur within 6-10 months.
  Assessment will be performed by calculating the time required to achieve complete retraction of the upper anterior teeth (six teeth) through clinical examination.
Change in the SNA angle | The cephalogram will be taken at three times: (T0) before the orthodontic treatment began, (T1) before the en-masse retraction began, (T3) at the end of the en-masse retraction phase (expected to occur within 6-10 months)
  This angle represents the position of the upper jaw in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
Change in the SNB angle | The cephalogram will be taken at three times: (T0) before the orthodontic treatment began, (T1) before the en-masse retraction began, (T3) at the end of the en-masse retraction phase (expected to occur within 6-10 months)
  This angle represents the position of the lower jaw in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken, and this angle will be measured in degrees.
Change in the ANB angle | The cephalogram will be taken at three times: (T0) before the orthodontic treatment began, (T1) before the en-masse retraction began, (T3) at the end of the en-masse retraction phase (expected to occur within 6-10 months)
  This angle represents the relationship between the upper and lower jaws in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken, and this angle will be measured in degrees.
Change in the SNPog angle | The cephalogram will be taken at three times: (T0) before the orthodontic treatment began, (T1) before the en-masse retraction began, (T3) at the end of the en-masse retraction phase (expected to occur within 6-10 months)
  This angle represents the position of the chin in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken, and this angle will be measured in degrees.
Change in the SN-GoMe angle | The cephalogram will be taken at three times: (T0) before the orthodontic treatment began, (T1) before the en-masse retraction began, (T3) at the end of the en-masse retraction phase (expected to occur within 6-10 months)
  This angle represents the position of the lower jaw in the cephalometric analysis in the vertical direction. Lateral cephalograms will be taken, and this angle will be measured in degrees.
Change in the MM angle | The cephalogram will be taken at three times: (T0) before the orthodontic treatment began, (T1) before the en-masse retraction began, (T3) at the end of the en-masse retraction phase (expected to occur within 6-10 months)
  This angle represents the amount of vertical divergence between the upper and lower jaws in the cephalometric analysis. Lateral cephalograms will be taken, and this angle will be measured in degrees.
Change in the Bjork's sum | The cephalogram will be taken at three times: (T0) before the orthodontic treatment began, (T1) before the en-masse retraction began, (T3) at the end of the en-masse retraction phase (expected to occur within 6-10 months)
  This angle represents the amount of vertical divergence in the cephalometric analysis. Lateral cephalograms will be taken, and this angle will be measured in degrees.
Change in Y-axis angle | The cephalogram will be taken at three times: (T0) before the orthodontic treatment began, (T1) before the en-masse retraction began, (T3) at the end of the en-masse retraction phase (expected to occur within 6-10 months)
  This angle represents the amount of vertical divergence in the cephalometric analysis. Lateral cephalograms will be taken, and this angle will be measured in degrees.
Change in the SN-U1 | The cephalogram will be taken at three times: (T0) before the orthodontic treatment began, (T1) before the en-masse retraction began, (T3) at the end of the en-masse retraction phase (expected to occur within 6-10 months)
  This angle represents the relationship of the upper anterior teeth with SN in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken, and this angle is going to be measured in degrees
Change in the GoMe-L1 angle | The cephalogram will be taken at three times: (T0) before the orthodontic treatment began, (T1) before the en-masse retraction began, (T3) at the end of the en-masse retraction phase (expected to occur within 6-10 months)
  This angle represents the relationship of the lower anterior teeth with the mandibular plane in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken, and this angle will be measured in degrees.
Change in the IIA angle | The cephalogram will be taken at three times: (T0) before the orthodontic treatment began, (T1) before the en-masse retraction began, (T3) at the end of the en-masse retraction phase (expected to occur within 6-10 months)
  This angle represents the relationship of the upper and lower anterior teeth in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken, and this angle is going to be measured in degrees.
Change in the SV-U1E distance | The cephalogram will be taken at three times: (T0) before the orthodontic treatment began, (T1) before the en-masse retraction began, (T3) at the end of the en-masse retraction phase (expected to occur within 6-10 months)
  This measurement represents the distance of the incisal edge of the maxillary incisors from the reference plane SV. Lateral cephalograms will be taken, and this measurement will be in millimeters.
Change in the SV-U1A distance | The cephalogram will be taken at three times: (T0) before the orthodontic treatment began, (T1) before the en-masse retraction began, (T3) at the end of the en-masse retraction phase (expected to occur within 6-10 months)
  This measurement represents the distance of the apex of the maxillary incisors from the reference plane SV. Lateral cephalograms will be taken, and this measurement will be in millimeters.
Change in the Nasolabial angle | The cephalogram will be taken at three times: (T0) before the orthodontic treatment began, (T1) before the en-masse retraction began, (T3) at the end of the en-masse retraction phase (expected to occur within 6-10 months)
  This angle represents the relationship of the upper lip with the nose in the cephalometric analysis. Lateral cephalograms will be taken, and this angle will be measured in degrees.
Change in the labiomental angle | The cephalogram will be taken at three times: (T0) before the orthodontic treatment began, (T1) before the en-masse retraction began, (T3) at the end of the en-masse retraction phase (expected to occur within 6-10 months)
  This angle represents the relationship of the lower lip with the chin in the cephalometric analysis. Lateral cephalograms will be taken, and this angle will be measured in degrees.
Change in the UL-E Line distance | The cephalogram will be taken at three times: (T0) before the orthodontic treatment began, (T1) before the en-masse retraction began, (T3) at the end of the en-masse retraction phase (expected to occur within 6-10 months)
  This measurement represents the relationship between the upper lip and the Ricketts line in cephalometric analysis. Lateral cephalograms will be taken, and this variable will be measured in mm.
Change in the LL-E Line distance | The cephalogram will be taken at three times: (T0) before the orthodontic treatment began, (T1) before the en-masse retraction began, (T3) at the end of the en-masse retraction phase (expected to occur within 6-10 months)
  This measurement represents the relationship between the Lower lip and the Ricketts line in cephalometric analysis. Lateral cephalograms will be taken, and this variable will be measured in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Younis Hajeer, DDS MSc PhD, Study Chair — Orthodontics Department, Faculty of Dentistry, University of Damascus
Locations (1):
- Department of Orthodontics, Faculty of Dentistry, University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spadari GS, Zaniboni E, Vedovello SA, Santamaria MP, do Amaral ME, Dos Santos GM, Esquisatto MA, Mendonca FA, Santamaria M Jr. Electrical stimulation enhances tissue reorganization during orthodontic tooth movement in rats. Clin Oral Investig. 2017 Jan;21(1):111-120. doi: 10.1007/s00784-016-1759-6. Epub 2016 Feb 26. PMID 26917494
- [Background] Davidovitch Z, Finkelson MD, Steigman S, Shanfeld JL, Montgomery PC, Korostoff E. Electric currents, bone remodeling, and orthodontic tooth movement. II. Increase in rate of tooth movement and periodontal cyclic nucleotide levels by combined force and electric current. Am J Orthod. 1980 Jan;77(1):33-47. doi: 10.1016/0002-9416(80)90222-5. PMID 6243448
- [Background] Shaadouh RI, Hajeer MY, Al-Sabbagh R, Alam MK, Mahmoud G, Idris G. A Novel Method to Accelerate Orthodontic Tooth Movement Using Low-Intensity Direct Electrical Current in Patients Requiring en-Masse Retraction of the Upper Anterior Teeth: A Preliminary Clinical Report. Cureus. 2023 May 24;15(5):e39438. doi: 10.7759/cureus.39438. eCollection 2023 May. PMID 37234453
- [Derived] Shaadouh RI, Hajeer MY, Alam MK, Sultan K, Aljabban O. Evaluation of the skeletal, dental, and soft-tissue changes after the en-masse retraction of upper anterior teeth stimulated by low-intensity electrical current: a randomized controlled clinical trial. BMC Oral Health. 2025 Jun 3;25(1):902. doi: 10.1186/s12903-025-06316-4. PMID 40462109